CLINICAL TRIAL: NCT06454526
Title: The Mindfulness Level of Manager Nurses, Leadership Behavior, Job Satisfaction, Job Performance, Burnout, Conflict Approach and Intention to Leave Will be Examined as Independent Variables.
Brief Title: Effects of Mindfulness-Based Program on Individual and Organizational Output of Frontline Manager Nurses:
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nazmiye Koseoglu, PhD student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022.275.IRB3.114
Record Dates: First submitted 2024-06-05; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Nurses; Mindfulness Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: All of the participants were blinded to the randomization procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): The group to which the 8-week Mindfulness-Based program will be applied.
  Interventions: Behavioral: Mindfulness Based Program
- Control (No Intervention): The group in which the 8-week Mindfulness-Based program will not be applied.

INTERVENTIONS:
Behavioral: Mindfulness Based Program — Mindfulness Based Program is an 8-week program with a total of 25 hours. The program, which consists of lectures, meditation and sharing areas, consists of the following topics: Six Senses and Pleasure, Mindfulness and Mind, Get Out of the Head and Enter the Body, Compassion, Meeting Challenges, Stress Reactions and Healing, Retreat Silence Day, Neuroplasticity and the Changing Brain and Wise Living.
  Arms: Experiment

SUMMARY:
The purpose of this randomized controlled study is to examine the effects of a mindfulness program applied to nurse managers on individual and organizational results. In the research, the Mindfulness-Based Program will be examined as the dependent variable, and the conscious awareness level of manager nurses, leadership behavior, job satisfaction, job performance, burnout, conflict approach and intention to leave will be examined as independent variables. The study was planned on the grounds that nurses need to be able to cope better with stress, reduce anxiety and burnout, and provide better job satisfaction in order to maintain a safe working life due to the increasing workload and difficulties of the healthcare system.

Hypotheses of the research are as follows:

H0: Mindfulness-Based Program is not effective on mindfulness, leadership behaviors, job satisfaction, job performance, burnout, conflict approach and intention to leave in manager nurses.

H1: Mindfulness-Based Program is effective on mindfulness, leadership behaviors, job satisfaction, job performance, burnout, conflict approach and intention to leave in manager nurses.

The population of the research will be all the responsible nurses working as low-level managers at Koç University Hospital and Kanuni Sultan Süleyman Training and Research Hospital. Responsible nurses who meet the sampling criteria and volunteer to participate in the study will be included in the study, and the participants will be randomly divided into intervention and control groups.

DETAILED DESCRIPTION:
In Turkey, studies on mindfulness in the nursing sample were carried out mostly descriptively, and nurses mindfulness levels were found to be at a medium level (Aşık and Albayrak, 2021; Özaydın, 2019). Considering the increasing workload and difficulties of the healthcare system, healthcare facility managers need to pay attention to the issue so that nurses can better cope with stress and reduce their anxiety and burnout in order to maintain a safe working life. This is a prerequisite for providing safe service to patients by providing better job satisfaction and performance. It may be possible to improve individual, team and organizational results with programs aimed at increasing the conscious awareness levels of manager nurses.

The purpose of this randomized controlled study is to examine the effects of a mindfulness program applied to nurse managers on individual and organizational results. In the research, the Mindfulness-Based Program will be examined as the dependent variable, and the conscious awareness level of manager nurses, leadership behavior, job satisfaction, job performance, burnout, conflict approach and intention to leave will be examined as independent variables. The study was planned on the grounds that nurses need to be able to cope better with stress, reduce anxiety and burnout, and provide better job satisfaction in order to maintain a safe working life due to the increasing workload and difficulties of the healthcare system.

Hypotheses of the research are as follows:

H0: Mindfulness-Based Program is not effective on mindfulness, leadership behaviors, job satisfaction, job performance, burnout, conflict approach and intention to leave in manager nurses.

H1: Mindfulness-Based Program is effective on mindfulness, leadership behaviors, job satisfaction, job performance, burnout, conflict approach and intention to leave in manager nurses.

The population of the research will be all the responsible nurses working as low-level managers at Koç University Hospital and Kanuni Sultan Süleyman Training and Research Hospital. Responsible nurses who meet the sampling criteria and volunteer to participate in the study will be included in the study, and the participants will be randomly divided into intervention and control groups.

The responsible nurses working at Koç University Hospital and Kanuni Sultan Süleyman Training and Research Hospital will be listed and the eligibility criteria for participation in the study (not having participated in the mindfulness program before) will be questioned. Participants included in the study will be listed and randomly divided into intervention and control groups. Randomization; Control and intervention groups will be assigned to the intervention or control group in the order of arrival, in line with the randomization list prepared in the Excel program using the random numbers method.

Before the implementation of the Mindfulness-Based Program , which will be implemented as an intervention in the research, all participants in the intervention and control groups were asked to use the Introductory Information Form, Conscious Awareness Scale, Minnesota Job Satisfaction Scale, Maslach Burnout Scale, Job Performance (Task/Contextual Performance) Scale, Rahim Organizational Conflict Inventory-2. Data (pretest) will be collected with (ROCI II) and the Intention to Leave Scale.

Conscious Awareness, job satisfaction, burnout, job performance and conflict inventory data will be collected again immediately (posttest) and three months later (follow-up) after the 8-week Mindfulness-Based Program implementation.

Data will be collected on charge nurses evaluations of leadership behaviors and intention to leave the subordinates they work with. For this purpose, the Introductory Information Form, Intention to Leave Scale and Leadership Behavior Scale were collected from the subordinates of the responsible nurses in the intervention and control group, before (pre-test), after (post-test) and three months later (follow-up) the intervention and control group. Data will be collected on a timely basis.

ELIGIBILITY:
Inclusion Criteria:

* Serving as a frontline nurse manager
* At least six months of managerial experience
* Not having participated in an eight-week Mindfulness-Based Program before

Exclusion Criteria:

* Serving as a lower-level manager for less than six months
* Having previously participated in an eight-week Mindfulness-Based Program

Termination Criteria:

* Participant withdraws from the study voluntarily.
* Participant's task change
* Participant leaving employment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | through study completion, an average of three months
  The Introductory Information Form, created by the researchers as a result of literature review, consists of 13 items. The content of the Form includes questions regarding sociodemographic (age, gender, educational status, marital status), professional characteristics (years of experience, management time, unit worked) and conscious awareness practices.
Conscious awareness scale (BIPÖ) | through study completion, an average of three months
  The Conscious Awareness Scale (BIPQ), developed by Brown and Ryan in 2003, was adapted into Turkish by Özyesil et al. in 2011. The scale consists of 15 items and is one-dimensional. The Likert-type scale is rated by participants on a scale of 1 to 6 (1: almost always, 6: almost never). As the total score obtained from the scale increases, the level of conscious awareness increases. A minimum of 15 and a maximum of 90 points are taken from the scale. An increase in the score obtained from the scale indicates that the level of conscious awareness is high.
Leadership Behavior Scale | through study completion, an average of three months
  The leadership behavior scale developed by Ekvall and Arvonen (1991) was adapted into Turkish by Tengilimoglu in 2005. The scale consists of 36 items and has 3 subscales. The Likert-type scale, which includes items expressing employee, task and change-oriented leadership behavior, is graded as (1) Strongly disagree, (2) Disagree, (3) Undecided, (4) Agree, (5) Strongly agree.
Minnesota Job Satisfaction Scale | through study completion, an average of three months
  Minnesota Job Satisfaction Scale, developed by Weiss, Dawis, England & Lofquist in 1967, was adapted into Turkish by Baycan (1985). The scale consists of three sub-dimensions: internal, external and general satisfaction and 20 items. It was made on a Likert type 5-point scale and was evaluated as (1) Very Dissatisfied, (2) Dissatisfied, (3) Undecided, (4) Satisfied, (5) Very Satisfied.
Maslach Burnout Scale | through study completion, an average of three months
  Maslach Burnout Scale, developed by Maslach and Jackson (1986), was adapted into Turkish by Ergin (1992). The scale consists of 22 items and evaluates burnout in three subscales (emotional exhaustion, depersonalization and personal accomplishment). A high score from the emotional exhaustion and depersonalization sub-dimensions of the scale and a low score from the personal success sub-dimension indicates that the level of burnout is high.
Job Performance (Task/Contextual Performance) Scale | through study completion, an average of three months
  The scale developed by Goodman and Svyantek (1999) was adapted into Turkish by Ünlü and Yürür in 2011. The scale, which includes 25 items, has two sub-dimensions: contextual performance and task performance. The scale is rated as a five-point Likert, "Definitely True-5 points" and "Definitely Not True-1 point".
Rahim Organizational Conflict Inventory-2 (ROCI II) | through study completion, an average of three months
  "The Rahim Organizational Conflict Inventory II-ROCI II" developed by Rahim (1983) was adapted into Turkish by Kozan and Ergin (1999). The five-point Likert type scale ((1) Strongly disagree, (2) Disagree, (3) Undecided, (4) Agree, (5) Strongly agree) consists of 31 items in total. Conflict management approaches have five sub-dimensions: Integrating, Compromising, Dominating, Avoiding, and Compromising.
Intention to Leave Scale | through study completion, an average of three months
  The Intention to Leave Scale, developed by Mobley, Horner and Hollingsworth (1978), was adapted into Turkish by Örücü and Özafşarlıoğlu (2013). The five-point Likert scale ((1) Strongly disagree, (2) Disagree, (3) Undecided, (4) Agree, (5) Strongly agree) type consists of 3 items and has no sub-dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Nazmiye Koseoglu, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa Graduate Education Institute, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghawadra SF, Abdullah KL, Choo WY, Phang CK. Mindfulness-based stress reduction for psychological distress among nurses: A systematic review. J Clin Nurs. 2019 Nov;28(21-22):3747-3758. doi: 10.1111/jocn.14987. Epub 2019 Jul 22. PMID 31267619
- [Result] Cummings GG, Tate K, Lee S, Wong CA, Paananen T, Micaroni SPM, Chatterjee GE. Leadership styles and outcome patterns for the nursing workforce and work environment: A systematic review. Int J Nurs Stud. 2018 Sep;85:19-60. doi: 10.1016/j.ijnurstu.2018.04.016. Epub 2018 May 3. PMID 29807190
- [Result] Janssen M, Heerkens Y, Kuijer W, van der Heijden B, Engels J. Effects of Mindfulness-Based Stress Reduction on employees' mental health: A systematic review. PLoS One. 2018 Jan 24;13(1):e0191332. doi: 10.1371/journal.pone.0191332. eCollection 2018. PMID 29364935
- [Result] Wong CA, Cummings GG, Ducharme L. The relationship between nursing leadership and patient outcomes: a systematic review update. J Nurs Manag. 2013 Jul;21(5):709-24. doi: 10.1111/jonm.12116. PMID 23865924
- See also: Cultivating leadership Dharma: Measuring the impact of regular mindfulness practice on creativity, resilience, tolerance for ambiguity, anxiety and stress. Journal of Management Development. — https://doi.org/10.1108/JMD-09-2015-0127